CLINICAL TRIAL: NCT05355909
Title: Effect of a Two Week Prehabilitation Program Before Major Abdominal Surgery
Brief Title: High Intensity PreHab Before Major Abdominal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PreHab in abdominal Surgery
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Prehabilitation
Keywords: ventilatory anaerobic threshold, Prehabilitation

STUDY DESIGN:
Intervention Model Description: Prospective, randomised, single blinded (patient-blinded) with two study groups
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- controll group (No Intervention): Standard of care without preoperative fitness program
- Interventional group (Experimental): After randomisation the patients will obtain a two week personalised fitness program to improve the preoperative fitness
  Interventions: Procedure: Individualized high intensity preoperative fitness training

INTERVENTIONS:
Procedure: Individualized high intensity preoperative fitness training — The individualised training program consists of stamina training, interval training and strength training. The personalised fitness training will be designed based on the FITT-VP (frequency, intensity, time, type, volume, progression) of the American College of Sports Medicine (ACSM) and will contain 6 training session within 2 weeks under supervision of professional sport physicians.
  Arms: Interventional group

SUMMARY:
The risk for major cardiac cardiovascular events (MACE) within the first 30 day after surgery is nit only associated to the patient relate risk factors but also to the kind of surgery. Surgical interventions can be distinguished infield risk (MACE <1%), moderate risk (MACE 1-5%) and high risk (MACE > 5%). In addition with patient related risk factors it can raise to values of 40%.

The preoperative aerobic fitness [oxygen uptake (VO2) at the ventilatory anaerobic threshold (VAT) <11 mL/kg/min] has been shown of particularly interest in identifying patients at increased risk of postoperative complications. In the last decade major interest was put in the question whether a preoperative personalised physical training may have beneficial effect on the preoperative fitness and on the occurrence of postoperative complications. In some small studies this benefit has been shown for abdominal and thoracic surgery.

However some of those studies are controversially discussed because of missing randomisation and methodical issues. Also most of the studies needs a four week training period. This may lead to ethical and logostical problems oncologic patients.

The aim of this study is to assess the effect of a personalised, high intensity trains program of two weeks on the preoperative fitness.

DETAILED DESCRIPTION:
The risk for major cardiac cardiovascular events (MACE) within the first 30 day after surgery is nit only associated to the patient relate risk factors but also to the kind of surgery. Surgical interventions can be distinguished infield risk (MACE <1%), moderate risk (MACE 1-5%) and high risk (MACE > 5%). In addition with patient related risk factors it can raise to values of 40%.

The preoperative aerobic fitness [oxygen uptake (VO2) at the ventilatory anaerobic threshold (VAT) <11 mL/kg/min] has been shown of particularly interest in identifying patients at increased risk of postoperative complications. In the last decade major interest was put in the question whether a preoperative personalised physical training may have beneficial effect on the preoperative fitness and on the occurrence of postoperative complications. In some small studies this benefit has been shown for abdominal and thoracic surgery.

However some of those studies are controversially discussed because of missing randomisation and methodical issues. Also most of the studies needs a four week training period. This may lead to ethical and logostical problems oncologic patients.

The aim of this study is to assess the effect of a personalised, high intensity trains program of two weeks on the preoperative fitness.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* BMI 18 - 35kg/m2
* Signed informed consent
* Elective abdominal surgery with moderate to high risk

Exclusion Criteria:

* Pregnancy of lactation
* Major trauma or massive haemorrhage with the last two weeks
* Inclusion of the patient in a interventional study
* Contraindication for preoperative fitness training or ergometry
* Transplantation surgery

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Preoperative fitness based on [oxygen uptake (VO2) at the ventilatory anaerobic threshold (VAT) <11 mL/kg/min] | 2 weeks
  (VO2) at the ventilatory anaerobic threshold (VAT) <11 mL/kg/min] between inclusion and end of personalised training hervor surgery.

SECONDARY OUTCOMES:
Quality of Life 36 (QoL-36) describes the quality of life of the patient with a scale ranging from 0 (worst outcome) to 100 (best outcome) between randomisation and end of training hervor surgery | 2 weeks
  Difference in Quality of Life 36 (QoL-36) describes the quality of life of the patient with a scale ranging from 0 (worst outcome) to 100 (best outcome) between randomisation and end of training hervor surgery

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Raab, MD, Principal Investigator — Medical University Innsbruck, Departement of Anaesthesiology and Intensive Care
Locations (1):
- Medical University Hospital, Innsbruck, Tyrol, Austria